CLINICAL TRIAL: NCT01361659
Title: Shockwave Treatment for Advanced Angina in Maastricht (SWAAM-study).
Brief Title: Shockwave Treatment for Advanced Angina in Maastricht
Acronym: SWAAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Medispec ltd. (Unknown)
Responsible Party: Prof Dr Harry Crijns, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-2-008
Record Dates: First submitted 2011-04-12; First posted 2011-05-27 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Angina
Keywords: anginal complaints; Lithotripsy; no option patients
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: shockwave treatment — 9 treatments in 3 months

SUMMARY:
There is an increasing number of patients with a coronary anatomy that does not allow additional revascularization procedures, while the patients suffer from angina pectoris at rest or at minimal exercise levels despite optimised medical therapy. There is a lack of therapeutic options for this group of so called "no-option patients". Goal of the project is to implement the shockwave therapy for no-option coronary artery disease patients and to evaluate its potential benefit on regional myocardial perfusion, on regional myocardial function and on the potential improvement in symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Chronic angina pectoris CCS (Canadian Cardiological Society) III or IV with documented reversible ischemia and/or hibernation.
* Patients demonstrates exercise tolerance test (ETT) duration < 10 minutes on a modified Bruce protocol
* No possibility of traditional revascularization by coronary artery bypass grafting (CABG) or Percutaneous coronary intervention (PCI)
* Patient's conditions stable for at least 3 months
* Life expectancy of > 12 months.

Exclusion Criteria:

* Unstable angina pectoris
* Haemodynamically significant valvular heart disease
* Myocardial infarction <3 month prior randomization
* Evidence of intracardiac thrombus
* Contraindication for Magnetic resonance imaging (MRI) (pacemaker, metallic prostheses)
* Patient is simultaneously participating in another device or drug study, or has participated in any clinical trial involving an experimental device or drug, including other drugs or devices enhancing cardiac neovascularization or any Extracorporeal Shock Wave Therapy (ESWT) machine for neovascularization of a competitor company within 3 months of entry into the study.
* Patients who are unwilling or unable to cooperate with the study procedure.
* Age < 18 years
* Cardiac or pulmonary malignancy
* No informed consent
* Known depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-05; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of exercise tolerance | after 6 months
  Modified Bruce protocol, changes compared to the baseline

SECONDARY OUTCOMES:
Improvement of myocardial perfusion | 6 months
  myocardial perfusion scintigraphy changes compared to the baseline
Number of Patients with Adverse Events as a Measure of Safety | 6 months
  Changes in electrocardiogram and cardiac enzymes (e.g. creatininekinase, troponin), clinical status and chestpain.
Improvement of quality of life | 6 months
  Number of anginal attacks/week, use of nitrates/week

CONTACTS AND LOCATIONS:
Overall Officials: H. Crijns, Prof Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands